CLINICAL TRIAL: NCT04811144
Title: Clinical Application of Er:YAG Dental Laser System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20170083
Record Dates: First submitted 2021-03-22; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Laser Therapy
Keywords: Er:YAG; dentistry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cavity group (Experimental): The 35 participants accepted Er:YAG laser treatment for dental cavity. Each participant was collected their data including history records, affected range check, X-ray&photo, treatment, pain index check, return visit check after two weeks by researchers.
  Interventions: Device: Er:YAG dental laser
- Sensitive Teeth group (Experimental): The 35 participants accepted Er:YAG laser treatment for sensitive teeth. Each participant was collected their data including history records, sensitive check, X-ray&photo, treatment, pain index and effectiveness check, return visit check after two weeks by researchers.
  Interventions: Device: Er:YAG dental laser
- Abnormal Frenum Attachment group (Experimental): The 35 participants accepted Er:YAG laser treatment for Abnormal Frenum Attachment. Each participant was collected their data including history records, abnormal position check, photo, cutting, pain index check, return visit check after three, five and seven days. by researchers.
  Interventions: Device: Er:YAG dental laser
- Peri-implantitis intervention group (Experimental): The 12 participants accepted Er:YAG laser treatment for Peri-implantitis. Each participant was collected their data including History records, measure periodontal pocket depth, anaerobes collect, X-ray, photo, CT, treatment, pain index check, return visit check after one week, two weeks, four weeks and three months, and six month check the effectiveness and collect anaerobes during every return visit. In the last return visit, X-ray and CT would be included
  Interventions: Device: Er:YAG dental laser
- Peri-implantitis control group (No Intervention): The 12 participants accepted mechanical debridement for Peri-implantitis. Each participant was collected their data including History records, measure periodontal pocket depth, anaerobes collect, X-ray, photo, CT, treatment, pain index check, return visit check after one week, two weeks, four weeks and three months, and six month check the effectiveness and collect anaerobes during every return visit. In the last return visit, X-ray and CT would be included

INTERVENTIONS:
Device: Er:YAG dental laser — To treat Cavity, Sensitive Teeth, Abnormal Frenum Attachment and Peri-implantitis by using Er:YAG Dental Laser system which manufactured by LightMed Dental Technology Corp
  Arms: Abnormal Frenum Attachment group; Cavity group; Peri-implantitis intervention group; Sensitive Teeth group

SUMMARY:
The study aim was to evaluate the effectiveness of Er:YAG dental laser treatment modality for cavity, sensitive teeth, abnormal frenum attachment and peri-implantitis.

DETAILED DESCRIPTION:
There are four indications will be included in this plan. They are Cavity, Sensitive Teeth, Abnormal Frenum Attachment and Peri-implantitis. Each indication has different procedures which are listed as below:

Cavity: history records, affected range check, X-ray&photo, treatment, pain index check, return visit check after two weeks. Sensitive Teeth: history records, sensitive check, X-ray&photo, treatment, pain index and effectiveness check, return visit check after two weeks. Abnormal Frenum Attachment: history records, abnormal position check, photo, cutting, pain index check, return visit check after three, five and seven days. Peri-implantitis: History records, measure periodontal pocket depth, anaerobes collect, X-ray, photo, CT, treatment, pain index check, return visit check after one week, two weeks, four weeks and three months, six months check the effectiveness and collect anaerobes during every return visit. In the last return visit, X-ray and CT would be included.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 20 years and above。
* Patients are available for multiple follow-up visits for the duration of the study.
* Having the mental ability to express informed consent.
* Patients clinically diagnosed as having Cavity, Sensitive Teeth, Abnormal Frenum Attachment or Peri-implantitis.

Exclusion Criteria:

* Severe diabetes and chronic diseases are excluded.
* CVA patients or the patients taking anti-rejection medicine and osteoporosis drugs for long-term should be excluded.
* Patient who suffer from photodermatosis and photosensitive patients (photoallergic).
* The health condition is not well after health education and physical therapy are excluded.
* Surgery on patients with serious diseases of the hemopoietic system (such as haemophilia and leukaemia).
* Malignant tumours, obligate precancerous tumours, hemangiomas.
* Coronary heart disease and chronic obstructive pulmonary diseases are excluded.
* Pregnant woman.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
pain index | two weeks
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is based solely on the ability to perform activities of daily living (ADLs) and can be used for adults and children 10 years old or older
sensitive check | two weeks
  The dentist asked participants few questions about dental status. Do you feel sudden discomfort in your teeth when you drink hot or cold beverages you once considered normal?
Abnormal Frenum Attachment | a week
  wound healing status
Probing depth | six months
  dentist measurement participant's probing depth the distance from the gingival margin to pocket base

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No